CLINICAL TRIAL: NCT06021444
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Pivotal, Non-inferiority Clinical Study to Evaluate the Efficacy and Safety of 'DKM420' in Knee Osteoarthritis Patients.
Brief Title: Efficacy and Safety of DKM420 in Patients With Osteoarthritis of Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKM-420-MD-1
Record Dates: First submitted 2023-04-17; First posted 2023-09-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 1:1 Parallel.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: 1. Blind: Investigator
  2. Un-blind: Investigator(or CRC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKM420 (Experimental): Injecting to one side knee.
  Interventions: Device: DKM420
- Conjuran (Active Comparator): Injecting to one side knee.
  Interventions: Device: Conjuran

INTERVENTIONS:
Device: DKM420 — A total of 3 doses will be applied at a dose of 2 mL over 3 weeks.
  Arms: DKM420
Device: Conjuran — A total of 3 doses will be applied at a dose of 2 mL over 3 weeks.
  Arms: Conjuran

SUMMARY:
To prove the non-inferiority of DKM420 by evaluating the injecting efficacy and safety DKM 420 and control for patients who have osteoarthritis of Knee.

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, active-controlled, pivotal, non-inferiority clinical study

ELIGIBILITY:
Inclusion Criteria:

* Men and Women who is over 40 under 80 ages.
* Diagnosed as osteoarthritis of Knee and satisfies the 3 of 6 ACR(American College of Rheumatology) conditions.
* Kellgren Lawrence grade (Ⅰ~Ⅲ) at Visit 1 or within 24 weeks.
* 100mm VAS(Visual Analogue Scale) over 40mm.
* Etc.

Exclusion Criteria:

- Pregnancy and lactating women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
100mm VAS(Visual Analogue Scale) | 16 weeks
  Change(The minimum value is 0mm, the maximum value is 100m, the lower the better.)

SECONDARY OUTCOMES:
100mm VAS(Visual Analogue Scale) | 2, 8 weeks
  Change(The minimum value is 0mm, the maximum value is 100m, the lower the better.)
K-WOMAC(Korean Western Ontario and McMaster Universities) | 2, 8, 16 weeks
  Change(Score from 0 to 96, the lower the better.)

CONTACTS AND LOCATIONS:
Locations (1):
- chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No